CLINICAL TRIAL: NCT01723813
Title: Phase I/II Study of Peptide Vaccination Associated With GM-CT-01, a Galactomannan Oligomer That Inhibits Galectin-3, in Patients With Advanced Metastatic Melanoma
Brief Title: Peptide Vaccinations Plus GM-CT-01 in Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to end of validity of peptide vaccine
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUC 10-001
Record Dates: First submitted 2012-09-28; First posted 2012-11-08 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Melanoma
Keywords: Immunotherapy; Tumor-specific peptides; GM-CT-01
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 : peptides + GM-CT-01 IV (Experimental): Tumor specific peptides: MAGE-3.A1 and / or NA17.A2 plus Galectin-3 inhibitor: GM-CT-01 systemic injections
  Interventions: Biological: Tumor specific peptides: MAGE-3.A1 and / or NA17.A2; Biological: Galectin-3 inhibitor: GM-CT-01 systemic injections
- Group 2 : peptides + GM-CT-01 IV+PT (Experimental): Tumor specific peptides: MAGE-3.A1 and / or NA17.A2 plus Galectin-3 inhibitor: GM-CT-01 systemic injections and Galectin-3 inhibitor: GM-CT-01 Peri-tumoral administration
  Interventions: Biological: Tumor specific peptides: MAGE-3.A1 and / or NA17.A2; Biological: Galectin-3 inhibitor: GM-CT-01 systemic injections; Biological: Galectin-3 inhibitor: GM-CT-01 Peri-tumoral administration

INTERVENTIONS:
Biological: Tumor specific peptides: MAGE-3.A1 and / or NA17.A2 — Each peptide will be given at a dose of 300 µg in 1 ml of sodium chloride 0.9%, every 3 weeks on 6 occasions, and will be administered at one site in arm or thigh, 20% of the dose intradermally and 80% of the dose subcutaneously.
Biological: Galectin-3 inhibitor: GM-CT-01 systemic injections — Systemic injection of GM-CT-01: GM-CT-01 will be administered by slow intravenous infusions at a dose of 280 mg/m2, on days +3, +6, +9, +12, +15, +18 after each of the 3rd, 4th, 5th and 6th vaccination.
Biological: Galectin-3 inhibitor: GM-CT-01 Peri-tumoral administration — GM-CT-01 will be injected peri-tumoral at a dose of 100 µg per tumor injected, on days +3, +6, +9, +12, +15, +18 after each of the 3rd, 4th, 5th and 6th vaccination. If a patient has one or two superficial metastases at day 43 of the treatment, one of these lesions will be treated. If a patient has more than two superficial metastases at day 43, two of these lesions will be treated.
  Arms: Group 2 : peptides + GM-CT-01 IV+PT

SUMMARY:
The purpose of this study is to determine whether the intravenous and/or GM-CT-01 administration can correct Tumor Infiltrating Lymphocytes (TIL) anergy and induce a more efficient and long-lasting anti-tumoral immune response following peptide vaccination.

DETAILED DESCRIPTION:
Human cancers express tumor antigens that can be targeted by cytolytic T lymphocytes (CTL). These antigens consist of a small peptide, derived from endogenous proteins, that is presented at the cancer cell's surface by an HLA class I molecule. Such antigenic peptides, including MAGE-3.A1 and NA17.A2, have been tested in experimental therapeutic vaccines to elicit CTL responses in cancer patients, mainly with metastatic melanoma. Up to now, only rare tumor responses have been observed.

Tumor resistance to CTL killing is the most likely explanation for the poor effectiveness of cancer vaccines. This resistance is probably acquired by the tumor during its development and selected by its repetitive challenge with spontaneous anti-tumoral immune responses. Recently, we have identified a novel mechanism causing anergy of tumor-associated T lymphocytes, and established new approaches to correct this anergy in vitro. Galectin-3, secreted by tumor cells, appears to inhibit CTL function the co-localization of the T cell receptor and the cluster of differentiation 8 coreceptor. Importantly, this functional defect is restored when anergic T cells are incubated with galectin-3 inhibitors such as the disaccharides lactose and N-acetyllactosamine, and the polysaccharide GM-CT-01. GM-CT-01 is a vegetal galactomannan oligomer, currently under clinical investigation in several types of solid malignancies for its capacity to inhibit galectins and to synergize with chemotherapy drugs.

Our observations suggest that treatment of cancer patients with GM-CT-01 could correct TIL anergy and induce a more efficient and long-lasting anti-tumoral immune response following peptide vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven cutaneous melanoma at one of the following American Joint Committee on Cancer stages : Regional metastatic disease (any T; N2c or N3; M0), no amenable to curative treatment by surgery or isolated limb perfusion.Distant metastatic disease (any T; any N; M1a, M1b or M1c*).*except uncontrolled brain metastasis and except Lactate dehydrogenase >1.5 upper normal value
* HLA-A1 or HLA-A2 (by serology or molecular biology)
* At least one of the two following conditions:

MAGE-3 gene expression by the tumor if patient is HLA-A1 NA17 gene expression by the tumor if patient is HLA-A2 (determined by reverse transcription and polymerase chain reaction amplification).

* Measurable Disease. Patients must have at least 1 measurable metastasis at study entry for all patients. In addition, patients candidates for enrollment in Group 2 who will receive peri-tumoral injections of GM-CT-01 must have at least 1 superficial metastasis (cutaneous, subcutaneous or superficial lymph node metastasis, with its largest diameter equal to or greater than 5, 5, or 10 mm, respectively) at study entry.
* Age ≥ 18 years.
* Karnofsky Performance status ≥70 or WHO performance status of 0 or 1
* Expected survival of at least 6 months.
* Laboratory values :

Platelet count ≥100x103/μL Leukocyte count ≥ 3x103/μL Hemoglobin ≥ 9 g/dL Aspartate transaminase and Alanine transaminase ≤ 2 times upper normal value Serum creatinine ≤1.5 times upper normal value Total bilirubin ≤ 1.5 times upper normal value Lactate dehydrogenase ≤ 1.5 times upper normal value

* Viral serology : negative antibodies for Hepatitis C Virus & HIV; negative antigens for Hepatitis B Virus.
* Patient should agree to perform biopsies and blood collections for translational research.
* Signed informed consent from the patient must be obtained.

Exclusion Criteria:

* Uncontrolled brain or central nervous system metastasis.
* Previous treatment for the melanoma within 6 weeks from inclusion, with any reagent known to modulate the immune system such as a cancer vaccine, interferon-alpha, interleukins or anti-CTLA-4 antibodies.
* Previous chemotherapy, radiotherapy, corticotherapy, or other immune suppressive therapy within 4 weeks from inclusion.
* Clinically significant cardiovascular disease (including cardiac insufficiency New York Heart Association grade III and IV, unstable angina, arrythmia, myocardial infarction, symptomatic congestive heart failure) in the past 12 months before enrollment.
* Other serious acute or chronic illnesses, e.g. active infections requiring antibiotics, bleeding disorders or other conditions requiring concurrent medications not allowed during this study.
* Other malignancy within 3 years prior to entry in the study, except for treated non-melanoma skin cancer and in situ cervical carcinoma.
* Active immunodeficiency disease or autoimmune disease (vitiligo is not an exclusion criterion).
* Lack of availability for immunological and clinical follow-up assessments.
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
* Subject pregnant or breastfeeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 30 days after last administration of Study drugs
  Change from baseline in adverse events will be recorded at each patient's visit and up to 30 days after last administration of study drugs. Measurements will use the Common Toxicity Criteria for Adverse Effects 4,0 scale
Response rate in both arms | Change from baseline at week 7 and week 20
  Efficacy of the combination of a peptide vaccine and GM-CT-01 injections measures performed by CT-scan or MRI

SECONDARY OUTCOMES:
Response rate in group 2 versus group 1 | Change from baseline at week 7 and week 20
  To determine whether addition of peri-tumoral injections of GM-CT-01 increase tumor response therefore response rate observed in group 1 will be compared with group 2
Time to Progression | From date of inclusion until the date of first documented progression or date of death from any cause, which ever came first, assessed up to 100 weeks
  patients will be followed every three months at consultation and with radiological examination, they will be assessed up to 100 weeks
Overall Survival | From day of inclusion to date of death
  patients will be followed every three months at consultation and with radiological examination, they will be assessed up to 100 weeks
Immunogenicity of the treatment | Change from baseline at week 20
  assessed at baseline and at week 20

OTHER OUTCOMES:
Translational research | baseline and at progression
  anti-tumoral immunological events in tumor samples obtained before and at progression
Pharmacokinetics of GM-CT-01 | Change from baseline at days 46 to 48
  serum concentration of GM-CT-01

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois BAURAIN, MD, PhD, Principal Investigator — Cliniques univeristaires Saint-Luc
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium